CLINICAL TRIAL: NCT02161744
Title: A Phase I Open- Label Study to Assess the Safety, Tolerability, and Preliminary Efficacy of a Single Intravenous Dose of Autologous Adipose Stem Cell (Adult Human) to Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Safety, Tolerability and Preliminary Efficacy of Adipose Derive Stem Cells for Patients With COPD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Arkansas Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICMS-2013-25
Record Dates: First submitted 2014-05-21; First posted 2014-06-12 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Adipose derived stem cells; Stromal vascular fraction cells; Pulmonary Function Tests; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Phase I open label study to assess safety and tolerability
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADSCs administration (Experimental): Patients with Chronic Obstructive Pulmonary Disease will be treated with a single dose of autologous adipose derived stem cells. Stem cells will be isolated using standard Lipoaspiration procedure under sterile conditions.
  Interventions: Biological: ADSCs administration

INTERVENTIONS:
Biological: ADSCs administration — 100- 240 cc of lipoaspirate will be extracted from the patient. The stromal vascular fraction (SVF) will be isolated with minimal manipulation. The cell pellet will be reconstituted in saline solution and administered intravenously to the patient.
  Other Names: Autologous Adipose Derived Stem Cells

SUMMARY:
The purpose of this study is: 1.- to assess the safety and tolerability of autologous adipose derived stem cells (aADSC) administered intravenously in patients with chronic obstructive pulmonary disease, and 2.- to assess if this therapy results in less decrease of lung function parameters (FEV1, FEV1/FVC and 6 min walking distance) compared with a control baseline of 6 weeks.

Patients will be followed up for 12 months after the therapy.

DETAILED DESCRIPTION:
STUDY DESIGN This is a Phase I open- label single-dose study in subjects with significant COPD. This is an expanded safety cohort. The investigators will enroll a minimum of 30 subjects. 6 week data of FEV1, FEV1/FVC, DLCO and 6 min walking distance values will be collected in all patients who are enrolled in the study (Baseline and 6 weeks after). Prior to the stem cell treatment, the patient will be assessed for 6 weeks by pulmonary function tests and 6 min walk tests. Then, patients will receive the infusion of stromal vascular fraction cells containing the aADSC (single intravenous dose). The standard therapy of COPD patients will not be interrupted during the duration of the study. Safety will be monitored on an ongoing basis, and an interim safety review will be conducted by the Investigator(s) and Sponsor after the first 20 patients have been enrolled and treated.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females ≥18 years.
2. Cognitive competitiveness.
3. Diagnosis of at least moderate COPD (postbronchodilator FEV1/FVC < 70% (<0.7), FEV1 < 80% predicted).
4. Diffusing capacity impairment (DLCO) assessed by single breath test (corrected for alveolar volume, 'DLVA').
5. Life expectancy greater than 12 months.
6. Ability to understand and provide signed informed consent, or have a designated legal guardian or spouse legally able and willing to make such decisions on the subject's behalf.
7. Reasonable expectation that patient will receive standard post-treatment care and attend all scheduled safety follow-up visits.
8. No changes in active pulmonary medications for heart failure during the two weeks prior enrollment.

10. Written informed consent. 11. Non-smoker or Past smoker, with 20 pack-years or more history

Exclusion Criteria:

1. Current smokers.
2. Unstable coronary disease.
3. Patients with industrial exposure to silica and/or asbestos or giant bullae.
4. Uncontrolled seizure disorder.
5. Dementia.
6. Presence of immune deficiency or autoimmune disease.
7. Alpha- 1 antitrypsin deficiency.
8. Cor pulmonale or diastolic heart failure NYHA class III or IV
9. Type 1 diabetes mellitus
10. Complicated type 2 diabetes mellitus.
11. Active tuberculosis or severe lung damage due to tuberculosis (extensive cavitation).
12. History of cancer within the past 5 years.
13. Clinically-significant hematologic, hepatic, or renal impairment as determined by screening clinical laboratory tests.
14. Systemic corticosteroids, cytostatics, immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), and DNA depleting or cytotoxic drugs taken within four weeks prior to study treatment.
15. Porphyria.
16. Allergy to sodium citrate or any "caine" type of local anesthetic.
17. Abnormal findings could include: known HIV infection or other immunodeficiency state, chronic active viral infection (such as hepatitis B or C), acute systemic infections (defined as patients undergoing treatment with antibiotics), gastrointestinal tract bleeding, or any severe or acute concomitant illness or injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Safety of adipose derived stem cells (ADSC) in Patient with COPD | 12 months
  Safety/tolerability of Adipose Derived Stem Cell (ADSC) in patients with Chronic Obstructive Pulmonary Disease (COPD) during the twelve-month study period as determined by the incidence and severity of of adverse events.

SECONDARY OUTCOMES:
Efficacy of ADSC in improving Shortness of Breath (SOB) | 2, 6 and 12 months
  The change (decrease) in patient Shortness Of Breath (SOB) as compared to baseline, measured in breath per minute, after administration of adipose derived stem cells (ADSC)
Efficacy of ADSC In Pulmonary Function Test (PFTs) | 2, 6, 12 months
  The change (improvement) in Pulmonary Function Test (PFTs) after administration of adipose derived stem cells (ADSC) as compared to baseline.
Efficacy of adipose derived stem cell in 6 MWT | 2, 6, 12 months
  Improvement in patient ability to walk as measure using a 6 minute walk test ( in meter) as compared to baseline
Efficacy of adipose derived stem cells in patient's perceived exertion. | 2, 6, 12 months
  The change from baseline in patient perceived exertion as measure using the modified BORG scale or Rate of perceive exertion (RPE) which ranges from 1(no perceived exertion at all) to 10 (maximum perceived exertion)
Efficacy in Quality of life using George's Respiratory Questionnaire | 2, 6, 12 months
  The change from baseline in patient quality of life as measure using the George's Respiratory Questionnaire
Efficacy in Quality of life using the Chronic Respiratory questionnaires | 2, 6, 12 months
  The change from baseline in patient quality of life as measure using the Chronic Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jason Holder, MD, Principal Investigator — Arkansas Heart Hospital
Locations (2):
- United States (2):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Arkansas Site Management Services LLC, Little Rock, Arkansas